CLINICAL TRIAL: NCT01597713
Title: A Trial Investigating the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of NNC0148-0000-0362 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN1954-3936; 2011-005147-27 (EudraCT Number); U1111-1125-2969 (Other: WHO)
Record Dates: First submitted 2012-05-10; First posted 2012-05-14 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2; Healthy
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part 1, level 1-7 escalating doses (Experimental)
  Interventions: Drug: NNC 0148-0000-0362; Drug: insulin glargine; Drug: placebo
- Part 2, cross-over (Experimental)
  Interventions: Drug: NNC 0148-0000-0362

INTERVENTIONS:
Drug: NNC 0148-0000-0362 — Subjects will be randomised to receive a single dose of NNC 0148-0000-0362 orally within each dose group
  Arms: Part 1, level 1-7 escalating doses
Drug: insulin glargine — As an active comparator, one standard dose will be given subcutaneously (s.c., under the skin) within each dose group
  Arms: Part 1, level 1-7 escalating doses
Drug: placebo — Subjects will receive a single dose of oral placebo within each dose group
  Arms: Part 1, level 1-7 escalating doses
Drug: NNC 0148-0000-0362 — Single low dose administered orally in randomised order on three dosing visits separated by a wash-out period
  Arms: Part 2, cross-over
Drug: NNC 0148-0000-0362 — Single high dose administered i.v. in randomised order on three dosing visits separated by a wash-out period
  Arms: Part 2, cross-over
Drug: NNC 0148-0000-0362 — Single high dose administered orally in randomised order on three dosing visits separated by a wash-out period
  Arms: Part 2, cross-over

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to investigate the safety, tolerability, pharmacokinetics (exposure of drug) and pharmacodynamics (effect of drug) of NNC 0148-0000-0362 as tablets in healthy volunteers.

The trial consists of two parts. In part 1, single escalating doses of NNC 0148-0000-0362, placebo or insulin glargine is given. In part 2, subjects will receive single doses of NNC 0148-0000-0362 administered orally or intravenously.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index 18-28 kg/m^2 (both inclusive)
* Subject who is considered to be healthy based on the medical history, physical examination, and the results of vital signs, electrocardiogram (ECG) and clinical laboratory tests performed during the screening visit, as judged by the investigator

Exclusion Criteria:

* Known or suspected hypersensitivity to trial products or related products
* Previous participation in this trial. Participation is defined as randomised
* Presence of clinically significant acute gastrointestinal symptoms (e.g. nausea, vomiting, heartburn or diarrhoea) within 2 weeks prior to dosing, as judged by the investigator
* Any chronic disorder or severe disease which, in the opinion of the investigator, might jeopardise subject's safety or compliance with the protocol

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 83 (Actual)
Dates: Start 2012-05; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | Recorded from trial product administration and until completion of Sub-visit G (i.e. Day 13) of the dosing visit

SECONDARY OUTCOMES:
Area under the serum insulin concentration-time curve (with Trial part 1) | From 0 to 288 hours after a single oral dose of NNC 0148-0000-0362 or a single subcutaneous (s.c.) dose of insulin glargine, respectively
Area under the glucose infusion rate (GIR)-time curve (Trial part 1) | From 0 to 24 hours after a single oral dose of NNC 0148-0000-0362 or a single s.c. dose of insulin glargine, respectively
Area under the serum insulin concentration-time curve (Trial part 2) | From 0 hours to infinity after a single dose of NNC 0148-0000-0362 administered orally as 1 and 3 tablets and intravenously, respectively

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Neuss, Germany

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com